CLINICAL TRIAL: NCT06805786
Title: Effect of Switching From Intermittently Scanned Continuous Glucose Monitoring to Real-time Continuous Glucose Monitoring on Glycemic Outcomes in Adults With Type 2 Diabetes
Brief Title: Effect of Switching From Intermittently Scanned to Real-time Continuous Glucose Monitoring on Diabetes Management in Adults With Type 2 Diabetes (Switch CGM T2D)
Acronym: Switch CGM T2D
Status: Recruiting | Type: Observational
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Switch CGM T2D
Record Dates: First submitted 2025-01-22; First posted 2025-02-03 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; continuous glucose monitoring; HbA1c; time in range
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (2):
- Real-time continuous glucose monitoring switch group (rtCGM switch group): adults with insulin-treated T2D that are switching from an isCGM to an rtCGM
  Interventions: Device: real-time continuous glucose monitor
- intermittently scanned continuous glucose monitoring group (isCGM group): adults with insulin-treated T2D that are remaining on an isCGM for the whole study

INTERVENTIONS:
Device: real-time continuous glucose monitor — Individuals who switched from using isCGM to rtCGM
  Groups: Real-time continuous glucose monitoring switch group (rtCGM switch group)

SUMMARY:
The goal of this prospective study is to evaluate diabetes outcomes and patient experience following a switch from second generation intermittently scanned continuous glucose monitor (isCGM) to real-time continuous glucose monitor (rtCGM) compared with participants with continued isCGM use among adults with insulin-treated type 2 diabetes (T2D) in a specialist endocrinology clinic setting in Canada. The study aims include:

Primary outcome - Evaluate change in percent time in range (TIR) at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with participants with continued second generation isCGM use.

Secondary outcomes - Compare glycemic and metabolic outcomes (ie. additional CGM metrics, HbA1c, and weight), and outcomes related to diabetes management (ie. self-reported hypoglycemia and change in total daily dose [TDD] of insulin) at 3-6 months follow-up in the rtCGM switch and isCGM cohorts among adults with insulin-treated T2D.

Exploratory outcomes - Evaluate patient-reported outcomes (PROs) in the rtCGM switch cohort only. PROs will include questions about device satisfaction and psychological distress at baseline and 3-6 months follow-up, and protocol-specific questions about Dexcom Care following use of the rtCGM device at 3-6 months follow-up. Additionally this study will compare percent TIR, percent TBR, percent TAR, and HbA1c between rtCGM switch and isCGM cohorts by insulin therapy subgroup (basal vs MDI therapy).

rtCGM switch participants will be enrolled at an LMC location and asked to complete PROs at baseline and 3-6 month follow-up. Continued isCGM participants will not be asked to complete PROs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Clinical diagnosis of T2D ≥ one year
* Using insulin for ≥ 6 months
* Continued FreeStyle Libre® 2 isCGM device (isCGM cohort) as of the study start date
* Would like to switch from a FreeStyle Libre® 2 isCGM device to a Dexcom® G7 rtCGM device (rtCGM switch cohort) as of the study start date
* Baseline HbA1c ≥ 7.5%
* Known rtCGM/isCGM start date (month and year)
* Exclusive use of isCGM for ≥ 3 months
* Data on LibreView platforms have percent sensor capture ≥ 70% for 14 days of available data up to 6 months prior to index date
* ≥ 1 value for TIR (%) up to 6 months (± 6 weeks) prior to index date
* ≥ 1 value for HbA1c (%) up to 6 months (± 6 weeks) prior to index date
* Data consent

Exclusion Criteria:

* Have a prior history of rtCGM within 12 months of the index date
* Recent or expectant change to antihyperglycemic medications or doses within 30 days of index date
* Recent or expectant titration of insulin dose ≥ 20% within 30 days of index date
* Are pregnant at the time of study enrollment or intending to become pregnant during the study
* Used the isCGM or rtCGM for < 3 months
* Using continuous subcutaneous insulin infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adults, who are active patients with insulin-treated T2D at LMC, who switch from a FreeStyle Libre® 2 device to a Dexcom® G7 (rtCGM switch cohort) or initiated a FreeStyle Libre® 2 and maintain isCGM use (isCGM cohort) after December 2024
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Percent Time in Range (TIR) | from enrollment to 6 months follow up
  evaluate change in percent TIR (3.9 to 10.0 mmol/L) at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with continued second generation isCGM cohort among propensity score matched cohorts of adults with insulin-treated T2D. Percent TIR will be reported from the patient's EMR or Clarity® and LibreView® platforms (last 14 days of available data closest to the index date or 6-month follow-up date, where percent sensor capture is ≥ 70%).

SECONDARY OUTCOMES:
Change in Percent Time Below Range (TBR) | from enrollment to 6 months follow up
  Evaluate change in percent TBR (<3.9 mmol/L) at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with continued second generation isCGM cohort among propensity score matched cohorts of adults with insulin-treated T2D.
Change In Percent Time Below Range (TBR) in Level 2 Hypoglycemia | from enrollment to 6 months follow up
  Evaluate change in percent TBR in level 2 hypoglycemia (<3.0 mmol/L) at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with continued second generation isCGM cohort among propensity score matched cohorts of adults with insulin-treated T2D.
Change in Percent Time Above Target Glucose Range (TAR) | from enrollment to 6 months follow up
  Evaluate change in percent TAR (>10.0 mmol/L) at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with continued second generation isCGM cohort among propensity score matched cohorts of adults with insulin-treated T2D.
Change in Mean Glucose | from enrollment to 6 months follow up
  Evaluate change in mean glucose (mmol/L) at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with continued second generation isCGM cohort among propensity score matched cohorts of adults with insulin-treated T2D.
Change in Glycemic Variability measured as Standard Deviation of Glucose (mmol/L) | from enrollment to 6 months follow up
  Evaluate change in glycemic variability reported as standard deviation (SD) (mmol/L) at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with continued second generation isCGM cohort among propensity score matched cohorts of adults with insulin-treated T2D.
Change in Glycemic Variability measured as the Coefficient of Variation of Glucose (%) | from enrollment to 6 months follow up
  Evaluate change in glycemic variability reported as CV (%) at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with continued second generation isCGM cohort among propensity score matched cohorts of adults with insulin-treated T2D.
Change in Frequency of Hypoglycemia Episodes | from enrollment to 6 months follow up
  Evaluate change in frequency of hypoglycemia episodes (frequency of events <3.9 mmol/L) at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with continued second generation isCGM cohort among propensity score matched cohorts of adults with insulin-treated T2D.
Percent Sensor Capture and Change in Percent Capture | from enrollment to 6 months follow up
  Evaluate Percent sensor capture and evaluate the change in percent sensor capture at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with continued second generation isCGM cohort among propensity score matched cohorts of adults with insulin-treated T2D.
Change in HbA1c | from enrollment to 6 months follow up
  Evaluate change in HbA1c (%) at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with continued second generation isCGM cohort among propensity score matched cohorts of adults with insulin-treated T2D.
Portion of Participants Achieving HbA1c ≤7.0% at Follow-Up | from enrollment to 6 months follow up
  Evaluate portion of participants achieving HbA1c ≤ 7.0% at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with continued second generation isCGM cohort among propensity score matched cohorts of adults with insulin-treated T2D.
Change in Weight | from enrollment to 6 months follow up
  Evaluate change in weight (kg) at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with continued second generation isCGM cohort among propensity score matched cohorts of adults with insulin-treated T2D.
Change in Weekly Incidence of Self-Reported Hypoglycemia | from enrollment to 6 months follow up
  Evaluate change in weekly incidence of self-reported hypoglycemia at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with continued second generation isCGM cohort among propensity score matched cohorts of adults with insulin-treated T2D.
Change in Proportion of Participants with ≥1 Self-reported Hypoglycemic Events per Week | from enrollment to 6 months follow up
  Evaluate change in proportion of participants with ≥1 self-reported hypoglycemic events per week at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with continued second generation isCGM cohort among propensity score matched cohorts of adults with insulin-treated T2D.
Change in Number of Non-Insulin Antihyperglycemic Agents (AHA) | from enrollment to 6 months follow up
  Evaluate change in number of non-insulin AHAs at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with continued second generation isCGM cohort among propensity score matched cohorts of adults with insulin-treated T2D.
Change in Total Daily Dose (TDD) of Insulin | from enrollment to 6 months follow up
  Evaluate change in total daily dose of insulin at 3-6 months follow-up after switching from a second generation isCGM system to a rtCGM system compared with continued second generation isCGM cohort among propensity score matched cohorts of adults with insulin-treated T2D.
Number of rtCGM Discontinuations | from enrollment to 6 months follow up
  Evaluate the number of rtCGM discontinuations at 3-6 months follow-up only for the cohort switching from a second generation isCGM system to a rtCGM system.

OTHER OUTCOMES:
Glucose Monitoring Device Satisfaction Scale (GMSS) | from enrollment to 6 months follow up
  includes questions about device satisfaction, filled out only by the cohort switching from isCGM to rtCGM
Diabetes Distress Scale (DDS) | from enrollment to 6 months follow up
  includes questions about psychological distress , filled out only by the cohort switching from isCGM to rtCGM
Protocol-Specific Dexcom Care Survey | assessed at 3-6 month follow-up
  includes protocol-specific questions about rtCGM device, filled out only by the cohort switching from isCGM to rtCGM

CONTACTS AND LOCATIONS:
Locations (1):
- LMC Diabetes & Endocrinology Ltd., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This is a real-world study using data retrieved from a national Diabetes Registry. IPD will not be shared.